CLINICAL TRIAL: NCT00184496
Title: Switching From Morphine to Methadone. A Clinical, Pharmacological and Pharmacogenetic Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPI 03/008
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cancer
Keywords: Analgesics, Opioid/pharmacokinetics; Humans; Methadone/therapeutic use; Neoplasms/complications; pain/drug therapy
MeSH Terms: conditions — Neoplasms | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- methadon (Active Comparator): Morphine methadone stop and go switch
  Interventions: Drug: Methadone
- Methadone (Active Comparator): Methadon morphine overlap switch
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — To methods for switching morphine to methadon. Stop-and go versus overlap

SUMMARY:
Cancer patients on morphine for chronic pain, with side effects or unsatisfactory pain relief, will be rotated to Methadone. We will try to find out what is the best methode to rotate, and the equivalent dosage.

DETAILED DESCRIPTION:
This study is based on the clinical observation that patients who are not well controlled on morphine or oxycodone may benefit from switching to another opioid, in this case methadone. Although the mechanism for such switch is not completely understood, evidence indicates that opioids with different chemical structures have different characteristics, not least in relation to new knowledge about genetic variation in opioid receptors. Another challenge is that there is much uncertainty regarding equianalgesic dose ratios for morphine and methadone. It seems that the higher the morphine doses, the relatively lower methadone doses are needed to substitute morphine. Furthermore, there is uncertainty to which switching procedures one should use, the most common ones are "stop and go" and a three days switch. Finally, it is reported that methadone may increase the QT interval of the ECG, and thus increase the risk for the ventricular arrhythmia Torsade de pointe. The aim of this randomized, open label, multicenter study is primarily to compare the switching procedures, but it will also provide more knowledge about equianalgesic dose ratios, the effect of methadone on the QT interval, genetical factors that may characterize patients needing opioid switch as well as their response to it, and finally if pharmacokinetic factors plays a role.

ELIGIBILITY:
Inclusion Criteria:

* • Malignant disease.

  * On morphine and in need of opioid rotation. (A patient in need of opioid rotation is defined as having insufficient pain control with or without unacceptable side effects from opioids).
  * Able to complete the planned assessment schedules.
  * Above 18 years of age.
  * If out-patient, the patient lives with someone who can observe him/her.
  * Given informed consent according to the ethical guidelines.

Exclusion Criteria:

* Not able to read or write in Norwegian
* The patient has participated in a clinical study 4 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The overall aim of the present study is to validate the switching procedure from morphine to methadone for patients with advanced cancer and a short life expectancy. More specifically, we will: | 2 weeks

SECONDARY OUTCOMES:
Collect blood samples for present and future genetic analyses in order to explore inter individual variations in methadone and morphine doses based upon possible polymorphisms. | 2 weeks
Compare the QT-intervals on electrocardiograms obtained before and after start with methadone. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD,PhD Prof., Principal Investigator — St Olavs University Hospital, Trondheim
Locations (1):
- St Olavs Hospital, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Moksnes K, Dale O, Rosland JH, Paulsen O, Klepstad P, Kaasa S. How to switch from morphine or oxycodone to methadone in cancer patients? a randomised clinical phase II trial. Eur J Cancer. 2011 Nov;47(16):2463-70. doi: 10.1016/j.ejca.2011.06.047. Epub 2011 Jul 19. PMID 21775131